CLINICAL TRIAL: NCT02622516
Title: Effectiveness of Additional Protocol Exercises for Cervical Mobility and Proprioception in Vestibular Rehabilitation: a Randomized Controlled Trial
Brief Title: Cervical Mobility and Vestibular Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Viviane de Souza Pinho Costa (Other)
Responsible Party: Sponsor-Investigator, Viviane de Souza Pinho Costa, Viviane, Universidade Norte do Paraná
Organization: Universidade Norte do Paraná (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Viviane-Unopar
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Vestibular Diseases
Keywords: Rehabilitation; Physical Therapy Specialty; Postural Balance; Vertigo; Dizziness
MeSH Terms: conditions — Vestibular Diseases; Vertigo; Dizziness | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (IG) (Active Comparator): Participants in the intervention group subjects (IG) will receive physiotherapy treatment in vestibular rehabilitation based on multisensory exercises consisting of the group of therapeutic proposals that stimulation of the vestibular, proprioceptive and visual associated with manual therapy treatment proposed by the techniques cervical global pompage and classic massage therapy on neck and shoulder girdle .
  Interventions: Other: Intervention Group (IG)
- Control Group (CG) (Experimental): Participants in the control group subjects (CG) will receive physiotherapy treatment in vestibular rehabilitation based on Cawthorne and Cooksey Exercises, consisting of eye movements in different directions, slowly and quickly; head movements in different planes, with open and closed eyes, slow and fast; and body exercises such as lifting and sit, walk open and closed eyes, up and down ramps and stairs, as well as some activities and ball games.
  Interventions: Other: Control Group (CG)

INTERVENTIONS:
Other: Intervention Group (IG) — Therapeutic approaches to this proposal are intended to promote muscle relaxation to increase range of motion and analgesia of neck and shoulder girdle region, as well as the fascial release these regions with the intervention of cervical global pompage, exercises for body mobility for upper limb and trunk in the positions supine, lateral and dorsal, sitting and standing and gradually followed by proprioceptive exercises to the lower limbs and trunk in sitting and standing positions with aid devices such as foams, pool baguettes, balance boards, Swiss balls, steps, trampolines and BOSU ( BOSU® Home Balance Trainer ).
  The exercises will be held in individual treatments lasting sixty minutes with a frequency of once a week for all group members.
  Other Names: Multisensory Exercises Protocol of Vestibular Rehabilitation
  Arms: Intervention Group (IG)
Other: Control Group (CG) — The exercises consist of eye movements in different directions, slow and fast; head movements in different planes, with open and closed eyes, slow and fast; and body exercises such as lifting and sit, walk open and closed eyes, up and down ramps and stairs, as well as some activities and ball games.
  The exercises will be held in individual treatments lasting sixty minutes with a frequency of once a week for all group members.
  Other Names: Conventional Protocol of Cawthorne & Cooksey Exercises
  Arms: Control Group (CG)

SUMMARY:
Vertigo, dizziness and imbalance are the main symptoms of vestibular dysfunction. They can lead to physical consequences, such as the reduction of postural control and falls, psychological and / or psychiatric consequences such as anxiety and depression, panic and cognitive changes, especially in the elderly. It is known that individuals affected by these disorders may improve with the completion of vestibular rehabilitation protocol.Treatment protocols can introduce variability of exercises to control the signs and symptoms related to vestibular diseases, in order to customize the treatment to affected individuals .

DETAILED DESCRIPTION:
The objective of this study will be to compare the effectiveness of a multisensory exercises protocol of vestibular rehabilitation versus conventional protocol of Cawthorne & Cooksey exercises for the treatment of patients with vestibular disorders. Methods: There will be a Clinical Trial Random, blind, Hidden Allocation. The sample will consist of 54 subjects submitted to two different protocols of vestibular rehabilitation exercises (Intervention Group (IG) and Control Group (CG)), to be held with individual treatment once a week, totaling 12 attendences. All will be assessed before and after treatment and the main variables analyzed are general characteristics of the clinical signs and symptoms caused by vestibular diseases, perception of quality of life and functional capacity paras activities of daily life, body flexibility, range of motion in the region cervical, parameters of static and dynamic postural balance and the perception of the results promoted by the treatment of vestibular rehabilitation and will compare the results of the groups. Expected results: It is expected, clinically, that subjects who receive treatment through multisensory exercises Protocol for VR present reduction of clinical signs and symptoms of dizziness, complaints of pains and cervical joint limitations, parameters of improvement related to postural balance, aspects of functional capacity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* People from the age of majority (18 years) to 69 years, considered by the population division in youth, adults and older people to 69 years according to the World Health Organization (WHO) , of both genders, with commitment by diagnosed peripheral vestibular disorders clinically by a doctor, including the peripheral vestibular type Benign Paroxysmal Positional Vertigo (BPPV), with vestibular symptoms, with higher scores than or equal to a spot on the Visual Analogue Scale (VAS) Dizziness or higher rank than or equal to 16 points in the questionnaire dizziness Handicap Inventory (DHI).

Exclusion Criteria:

* Elderly aged 70 or more, which have visual impairment and/or total hearing, orthopedic disorders that limit the realization of the proposed activities, nervous system injuries that cause damage engines and/or additional sensitive and diagnostics of Ménière's disease.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Balance Measure from force platform (COP Measure) | 12 weeks
  To assess postural control by means of a force platform named BIOMEC400 (EMG System Brazil, SP Ltda), and the data sampled at 100 Hz variables will be used: pressure downtown area (A-COP in cm2), average velocity of COP (VEL in cm/sec), amplitude (AMP cm) and average frequency of COP (FM in Hz) in both movement directions: anterior-posterior (A/P ) and medial-lateral (M/L).

SECONDARY OUTCOMES:
Timed Up and Go test (TUG) | 12 weeks
  Which evaluates the risk of falls. Starting from the sitting position, analyzes the transfer from sitting to standing, stability and progress of the ongoing changes without using compensatory strategies .
Functional Reach test (FRT) | 12 weeks
  Measure the mobility test with emphasis on the assessment of the balance. It is performed by asking the individual to stand up, next to a wall with shoulder flexion 90° and upper limbs in extension. Then he asks the individual to conduct an anterior flexion of the trunk, without the heels lose contact with the ground. Performance is measured by the distance traveled by the body's displacement (in centimeters), with the mean of three test attempts.
Agility Test | 12 weeks
  Agility test to evaluate the agility and dynamic balance.
Dizziness Handicap Inventory (DHI) | 12 weeks
  This questionnaire was developed and validated in order to evaluate the self- perception of the tax effects of dizziness on quality of life.
Vestibular Disorders Activities of Daily Living Scale Questionaire (VADL) | 12 weeks
  Evaluates the impact of dizziness and body imbalance in daily activities of vestibular individuals.
Visual Analog Scale (VAS) of Dizziness | 12 weeks
  Which indicates the intensity of vertigo symptoms, and varies on a numerical scale from zero to ten, where zero indicates the absence of dizziness and ten, the worst intensity of dizziness.
Fleximeter | 12 weeks
  Fleximeter to assess the range of motion of the cervical spine, consisting in a gravity - dependent inclinometer, whose range is a degree, attached to a velcro tape to be secured in head circumference participant.

CONTACTS AND LOCATIONS:
Overall Officials: Viviane SP Costa, Study Director — Universidade Norte do Paraná

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adamo DE, Pociask FD, Goldberg A. The contribution of head position, standing surface and vision to postural control in young adults. J Vestib Res. 2013;23(1):33-40. doi: 10.3233/VES-130473. PMID 23549053
- [Result] Albera R, Ciuffolotti R, Di Cicco M, De Benedittis G, Grazioli I, Melzi G, Mira E, Pallestrini E, Passali D, Serra A, Vicini C. Double-blind, randomized, multicenter study comparing the effect of betahistine and flunarizine on the dizziness handicap in patients with recurrent vestibular vertigo. Acta Otolaryngol. 2003 Jun;123(5):588-93. doi: 10.1080/00016480310001475. PMID 12875580
- [Result] Badke MB, Miedaner JA, Shea TA, Grove CR, Pyle GM. Effects of vestibular and balance rehabilitation on sensory organization and dizziness handicap. Ann Otol Rhinol Laryngol. 2005 Jan;114(1 Pt 1):48-54. doi: 10.1177/000348940511400109. PMID 15697162
- [Result] Ricci NA, Aratani MC, Caovilla HH, Cohen HS, Gananca FF. Evaluation of properties of the Vestibular Disorders Activities of Daily Living Scale (Brazilian version) in an elderly population. Braz J Phys Ther. 2014 Mar-Apr;18(2):174-82. doi: 10.1590/s1413-35552012005000144. Epub 2014 Mar 19. PMID 24676704
- [Result] Han BI, Song HS, Kim JS. Vestibular rehabilitation therapy: review of indications, mechanisms, and key exercises. J Clin Neurol. 2011 Dec;7(4):184-96. doi: 10.3988/jcn.2011.7.4.184. Epub 2011 Dec 29. PMID 22259614
- [Result] Meldrum D, Herdman S, Moloney R, Murray D, Duffy D, Malone K, French H, Hone S, Conroy R, McConn-Walsh R. Effectiveness of conventional versus virtual reality based vestibular rehabilitation in the treatment of dizziness, gait and balance impairment in adults with unilateral peripheral vestibular loss: a randomised controlled trial. BMC Ear Nose Throat Disord. 2012 Mar 26;12:3. doi: 10.1186/1472-6815-12-3. PMID 22449224
- [Result] da Silva RA, Bilodeau M, Parreira RB, Teixeira DC, Amorim CF. Age-related differences in time-limit performance and force platform-based balance measures during one-leg stance. J Electromyogr Kinesiol. 2013 Jun;23(3):634-9. doi: 10.1016/j.jelekin.2013.01.008. Epub 2013 Feb 10. PMID 23403137
- [Result] Horak FB. Postural compensation for vestibular loss and implications for rehabilitation. Restor Neurol Neurosci. 2010;28(1):57-68. doi: 10.3233/RNN-2010-0515. PMID 20086283